CLINICAL TRIAL: NCT02600858
Title: Exogenous Effects of Standard Medical Care (Dopamine) on Motor Learning of an Upper Limb Task in Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Lee Dibble, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IRB_00085073_UL
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Training "off" medication (Experimental): Participants will train on the upper limb feeding task before taking their first daily dose of standard dopamine medication for Parkinson's disease, i.e. while "off" dopamine replacement medication
  Interventions: Behavioral: Upper limb feeding training
- Training "on" medication (Other): Participants will train on the upper limb feeding task after taking their first daily dose of standard dopamine medication for Parkinson's disease, i.e. while "on" dopamine replacement medication
  Interventions: Behavioral: Upper limb feeding training

INTERVENTIONS:
Behavioral: Upper limb feeding training — Participants will spoon two raw kidney beans at a time from a center proximal "start" cup to three distal "target" cups positioned 16 cm away at 45°, 90° and 135° around the start cup as fast as possible using their non-dominant hand. Spooning two beans between the start cup and a target cup is considered one repetition; each trial will consist of 15 repetitions. Participants will perform 50 trials per day for 3 consecutive days.

SUMMARY:
The study determines whether standard medical care (dopamine) affects learning and retention of an upper limb feeding task in people with Parkinson's disease (PD) and whether training on the feeding task generalises to performance on an untrained upper limb buttoning task. Half the participants will train on the feeding task after they have taken their first dose of dopamine for the day (i.e. "on" medication state), while the other half will train on the same feeding task before taking their first daily dose of dopamine (i.e. "off" medication state).

DETAILED DESCRIPTION:
Parkinson disease (PD) is an age related neurodegenerative disorder with symptomatic declines in motor function due to a loss of dopaminergic neurons within the basal ganglia.

Ironically, treatment with exogenous dopamine-replacement medication (e.g. levodopa) may have positive effects on existing motor skills such as handwriting or walking, but may have detrimental effects on the learning of motor skills necessary for effective rehabilitation.

Although dopamine medications are routinely prescribed to replace lost dopamine in the sensorimotor areas of the striatum, they may actually be "overdosing" the associative striatum, a candidate neuroanatomical correlate for motor learning. To date, however, this 'overdose' hypothesis has not been widely tested, given that few studies of motor learning in PD have reported or controlled for whether individuals were tested "on" or "off" their dopamine replacement medication.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease confirmed by neurologist
* Hoehn and Yahr stages 1 to 3
* On a stable dose of antiparkinsonian medication for the past month and will continue on this regime for at least another subsequent month
* Walks unaided

Exclusion Criteria:

* Not taking dopamine replacement therapy
* With prior surgical management for PD (e.g. deep brain stimulation)
* With medication-resistant freezing of gait
* Significant cognitive impairment (Montreal Cognitive Assessment score <18)
* Unstable medical conditions
* Other neurological conditions
* Unable to follow instructions or safely complete the training tasks

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Task performance (response time) at initial retention, adjusted for baseline (first trial of acquisition on Day 3) | Day 8 (i.e. 48 hours after the last block of training)

SECONDARY OUTCOMES:
Immediate decrement (difference in response time between initial retention and the last trial of acquisition) in task performance, adjusted for baseline (first trial of acquisition) | Day 5, Day 8 (i.e. 48 hours after the last block of training)
Delayed decrement (difference in response time between delayed retention and the last trial of acquisition) in task performance, adjusted for baseline (first trial of acquisition) | Day 5, Day 15 (i.e. 9 hours after the last block of training)
Rate of improvement | Day 1 through Day 3
  Rate of improvement (c) modelled on the exponential decay function: y = a + be(exp[-x/c]), where a is the final trial time value that the exponential decay function approaches (ie, asymptote), b is the scale of the learning from the first trial time to the value a, x is the trial number, 1/c is the number of trials needed to obtain asymptote (ie, 1 - e-1).
Nine hole peg test score | Day 15 (i.e. 9 days after the last block of training)
  Time taken to complete the Nine Hole Peg Test at delayed retention, adjusted for baseline (Nine Hole Peg Test score at baseline, i.e. 3 days prior to the first block of training)
Buttoning task score | Day 15 (i.e. 9 days after the last block of training)
  Time taken to complete the Buttoning task at delayed retention, adjusted for baseline (Buttoning task score at baseline, i.e. 3 days prior to the first block of training)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Dibble, PhD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States